CLINICAL TRIAL: NCT03972709
Title: A Phase II, Multicenter, Randomized, Single-Masked, Sham-Controlled Study to Assess Safety, Tolerability, and Efficacy of Intravitreal Injections of FHTR2163 in Patients With Geographic Atrophy Secondary to Age-Related Macular Degeneration (GALLEGO)
Brief Title: A Study Assessing the Safety, Tolerability, and Efficacy of Galegenimab (FHTR2163) in Participants With Geographic Atrophy Secondary to Age-Related Macular Degeneration (AMD)
Acronym: GALLEGO
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The benefit to risk balance did not support further treatment with galegenimab (FHTR2163).
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GR40973
Record Dates: First submitted 2019-05-31; First posted 2019-06-04 (Actual); Results first posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Macular Degeneration, Age-Related; Geographic Atrophy
MeSH Terms: conditions — Macular Degeneration; Geographic Atrophy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Galegenimab Q4W (Experimental): Participants will receive galegenimab every 4 weeks (Q4W). After completing the study's last visit (Week 76), eligible participants will have the option to enroll in open-label extension study NCT04607148 (GR42558) and receive open-label galegenimab injections.
  Interventions: Drug: Galegenimab
- Sham Control Q4W (Sham Comparator): Participants will receive Sham-control Q4W. After completing the study's last visit (Week 76), eligible participants will have the option to enroll in open-label extension study NCT04607148 (GR42558) and receive open-label galegenimab injections.
  Interventions: Drug: Sham Control
- Galegenimab Q8W (Experimental): Participants will receive galegenimab every 8 weeks (Q8W). After completing the study's last visit (Week 76), eligible participants will have the option to enroll in open-label extension study NCT04607148 (GR42558) and receive open-label galegenimab injections.
  Interventions: Drug: Galegenimab
- Sham Control Q8W (Sham Comparator): Participants will receive Sham-control Q8W. After completing the study's last visit (Week 76), eligible participants will have the option to enroll in open-label extension study NCT04607148 (GR42558) and receive open-label galegenimab injections.
  Interventions: Drug: Sham Control

INTERVENTIONS:
Drug: Galegenimab — Intravitreal (ITV) injections of galegenimab
  Other Names: FHTR2163, RG6147
  Arms: Galegenimab Q4W; Galegenimab Q8W
Drug: Sham Control — Sham control
  Arms: Sham Control Q4W; Sham Control Q8W

SUMMARY:
This study will evaluate the safety, tolerability, and efficacy of intravitreal injections of galegenimab (FHTR2163) administered every 4 weeks (Q4W) or every 8 weeks (Q8W) for approximately 76 weeks in participants with geographic atrophy (GA) secondary to age-related macular degeneration (AMD) compared with sham control. After completing the study's last visit (Week 76), eligible participants will have the option to enroll in open-label extension study NCT04607148 (GR42558) and receive open-label galegenimab (FHTR2163) injections.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 60 years at time of signing Informed Consent Form;
* Visual acuity: best-corrected visual acuity (BCVA) letter score >/= 24 letters (Snellen equivalent of 20/320 or better). If the study eye BCVA letter score is >/= 69 letters (Snellen equivalent of 20/40 or better), the non-study eye must have a BCVA letter score of >/= 44 letters (Snellen equivalent of 20/125 or better);
* Well-demarcated area of GA secondary to AMD with no evidence of prior or active choroidal neovascularization (CNV) in either eye.

Exclusion Criteria:

Ocular Exclusion Criteria, Study Eye:

* History of vitrectomy surgery, submacular surgery, or any surgical intervention for AMD;
* Previous laser photocoagulation or ITV anti-vascular endothelial growth factor (anti-VEGF) for CNV, diabetic macular edema, retinal vein occlusion, or proliferative diabetic retinopathy.

Ocular Exclusion Criteria, Both Eyes:

* GA in either eye due to causes other than AMD;
* Active uveitis and/or vitritis (grade trace or above) in either eye;
* Active, infectious conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye;
* Retinal pigment epithelium (RPE) tear that involves the macula in either eye;
* Previous participation in interventional clinical trials for GA or dry AMD, except for vitamins and minerals, regardless of the route of administration (i.e., ocular or systemic) within the last 6 months.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 372 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2022-10-27 (Actual); Study Completion 2022-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (72):
- United States (72):
  - Arizona Retina and Vitreous Consultants, Phoenix, Arizona
  - Retina Associates Southwest PC, Tucson, Arizona
  - California Retina Consultants, Bakersfield, California
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - The Retina Partners, Encino, California
  - Retina Consultants of Orange County, Fullerton, California
  - Jules Stein Eye Institute/ UCLA, Los Angeles, California
  - Northern California Retina Vitreous Associates, Mountain View, California
  - Retina Consultants, San Diego, Poway, California
  - Retinal Consultants Med Group, Sacramento, California
  - W Coast Retina Med Group Inc, San Francisco, California
  - California Retina Consultants, Santa Barbara, California
  - California Retina Consultants - Santa Maria, Santa Maria, California
  - Bay Area Retina Associates, Walnut Creek, California
  - Retina Consultants of Southern Colorado PC, Colorado Springs, Colorado
  - Southwest Retina Consultants, Durango, Colorado
  - Colorado Retina Associates, PC, Lakewood, Colorado
  - Rand Eye, Deerfield Beach, Florida
  - Florida Eye Associates - Melbourne 2nd Office, Melbourne, Florida
  - Retina Specialty Institute, Pensacola, Florida
  - Retina Vitreous Assoc of FL, St. Petersburg, Florida
  - Southern Vitreoretinal Associates, Tallahassee, Florida
  - Southeast Retina Center, Augusta, Georgia
  - Georgia Retina PC, Marietta, Georgia
  - Illinois Eye and Ear Infirmary, Chicago, Illinois
  - University Retina and Macula Associates, PC, Oak Forest, Illinois
  - Wolfe Eye Clinic, West Des Moines, Iowa
  - Vitreo Retinal Consultants, Wichita, Kansas
  - Maine Eye Center, Portland, Maine
  - The Retina Care Center, Baltimore, Maryland
  - Johns Hopkins Hospital., Baltimore, Maryland
  - Retina Group of Washington, Chevy Chase, Maryland
  - Cumberland Valley Retina Consultants, Hagerstown, Maryland
  - Mass Eye and Ear Infirmary, Boston, Massachusetts
  - Vitreo-Retinal Associates, Grand Rapids, Michigan
  - Associated Retinal Consultants PC, Royal Oak, Michigan
  - VitreoRetinal Surgery, PLLC.; DBA Retina Consultants of Minnesota, Edina, Minnesota
  - Midwest Vision Research Foundation, Chesterfield, Missouri
  - The Retina Institute, St Louis, Missouri
  - Sierra Eye Associates, Reno, Nevada
  - Envision Ocular, LLC, Bloomfield, New Jersey
  - Mid Atlantic Retina, Cherry Hill, New Jersey
  - Retina Associates of NJ, Teaneck, New Jersey
  - Retina Vitreous Center, PA, Toms River, New Jersey
  - Long Is. Vitreoretinal Consult, Hauppauge, New York
  - Ophthalmic Consultants of Long Island, Oceanside, New York
  - Retina Associates of Western New York, Rochester, New York
  - The Retina Consultants, Slingerlands, New York
  - Western Carolina Retinal Associate PA, Asheville, North Carolina
  - Charlotte Eye Ear Nose and Throat Associates PA, Charlotte, North Carolina
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Retina Assoc of Cleveland Inc, Cleveland, Ohio
  - Cleveland Clinic Foundation; Cole Eye Institute, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Retina Associates of Cleveland - Middleburg Heights Location, Middleburg Heights, Ohio
  - Retina Associates of Cleveland - Youngstown Location, Youngstown, Ohio
  - Casey Eye Institute, Portland, Oregon
  - Mid Atlantic Retina - Wills Eye Hospital, Philadelphia, Pennsylvania
  - Palmetto Retina Center, West Columbia, South Carolina
  - Southeastern Retina Associates Chattanooga, Chattanooga, Tennessee
  - Charles Retina Institute, Germantown, Tennessee
  - Tennessee Retina PC, Nashville, Tennessee
  - Retina Res Institute of Texas, Abilene, Texas
  - Austin Retina Associates, Austin, Texas
  - Austin Clinical Research LLC, Austin, Texas
  - Retina Foundation of the Southwest, Dallas, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas
  - Retina Consultants of Texas, The Woodlands, Texas
  - Retina Consultants of Houston, The Woodlands, Texas
  - Rocky Mountain Retina, Salt Lake City, Utah
  - Spokane Eye Clinical Research, Spokane, Washington
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

RESULTS

PARTICIPANT FLOW:
Groups:
- All Sham: Participants will receive Sham-control Q4W or Q8W. After completing the study's last visit (Week 76), eligible participants will have the option to enroll in open-label extension study NCT04607148 (GR42558) and receive open-label galegenimab injections.
Period: Overall Study
Arm/Group | Galegenimab Q4W | Galegenimab Q8W | All Sham
Started | 149 | 75 | 148
Completed | 67 | 35 | 72
Not Completed | 82 | 40 | 76
Not completed — Withdrawal by Subject | 18 | 7 | 14
Not completed — Study Terminated by Sponsor | 48 | 25 | 50
Not completed — Physician Decision | 1 | 0 | 0
Not completed — COVID-19 | 0 | 1 | 1
Not completed — Lost to Follow-up | 6 | 1 | 2
Not completed — Death | 5 | 1 | 4
Not completed — Adverse Event | 3 | 1 | 4
Not completed — Subject Expired Due to SAE with Onset Beyond Protocol Reporting Period | 0 | 1 | 0
Not completed — Subject in Nursing Home, Unable to Attend Visit | 0 | 0 | 1
Not completed — Subject Unable to be Contacted | 0 | 1 | 0
Not completed — Subject Discontinuation Due to AEs with Onset Beyond Study Reporting Period | 0 | 1 | 0
Not completed — Subject Moved | 0 | 1 | 0
Not completed — Missed Study Visits | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Galegenimab Q4W | Galegenimab Q8W | All Sham | Total
Number analyzed (Participants) | 149 | 75 | 148 | 372
Age, Continuous [Mean (Standard Deviation); unit: Years] | 78.9 (7.3) | 78.4 (7.8) | 78.0 (7.7) | 78.4 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 50 | 83 | 222
  Male | 60 | 25 | 65 | 150
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 3 | 10
  Not Hispanic or Latino | 143 | 71 | 145 | 359
  Unknown or Not Reported | 3 | 0 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 147 | 74 | 146 | 367
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Geographic Atrophy (GA) Area From Baseline to Week 72 as Measured by Fundus Autofluorescence (FAF)
Description: GA is an advanced stage of age-related macular degeneration (AMD) and is characterized by loss of photoreceptors, retinal pigment epithelium, and choriocapillaris. In the early stages of GA, patients typically show minimal changes in central visual acuity although patients often still experience significant symptoms from visual dysfunction, such as reduced contrast sensitivity, and a decrease in reading speed. In the later stages, as the GA lesion expands into the fovea, a profound decrease in central visual acuity occurs with a decline in activities of daily living. The change in GA lesion area was measured by FAF and analysis of FAF images was performed by the central reading center. A positive change from baseline indicates an increase in size of GA lesion area (worsening; disease progression).
Time Frame: Baseline, Week 72
Population: Modified intent-to-treat (mITT) population includes all randomized patients who received at least one dose of study drug, and have a baseline measurement and at least one post-baseline measurement of GA area by FAF, subjects grouped according to treatment assigned at randomization. Participants analyzed in this outcome measure were those included in mixed models for repeated measures (MMRM) analysis.
Measure: Mean (Standard Error); unit: mm^2
Arm/Group | Galegenimab Q4W | Galegenimab Q8W | All Sham
Number analyzed (Participants) | 138 | 67 | 132
mm^2 | 2.60 (0.133) | 2.43 (0.189) | 2.31 (0.133)
Statistical Analysis 1: Comparison: Galegenimab Q4W vs All Sham; Test type: Superiority; p = 0.1206, MMRM; Difference in Adjusted Means = 0.29, 95% CI [-0.08 to 0.66], Standard Error of Mean 0.188
Statistical Analysis 2: Comparison: Galegenimab Q8W vs All Sham; Test type: Superiority; p = 0.6127, MMRM; Difference in Adjusted Means = 0.12, 95% CI [-0.34 to 0.57], Standard Error of Mean 0.231

2. Secondary Outcome: Percentage of Participants With Ocular Adverse Events in the Study Eye
Description: An AE was defined as any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether considered related to the medicinal product, any new disease or exacerbation of an existing disease, recurrence of an intermittent medical condition, or any deterioration in a laboratory value or other clinical test. Ocular AEs are the events which are localized in the ocular region.
Time Frame: From baseline to Week 76
Population: Safety analysis population included all randomized participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Galegenimab Q4W | Galegenimab Q8W | All Sham
Number analyzed (Participants) | 149 | 75 | 148
percentage of participants | 49.7 | 48 | 32.4

3. Secondary Outcome: Percentage of Participants With Ocular Adverse Events in the Fellow Eye
Description: as for outcome 2
Time Frame: From baseline to Week 76
Population: Safety analysis population included all randomized participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Galegenimab Q4W | Galegenimab Q8W | All Sham
Number analyzed (Participants) | 149 | 75 | 148
percentage of participants | 29.5 | 20.0 | 22.3

4. Secondary Outcome: Percentage of Participants With Systemic Adverse Events
Description: An AE was defined as any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether considered related to the medicinal product, any new disease or exacerbation of an existing disease, recurrence of an intermittent medical condition, or any deterioration in a laboratory value or other clinical test. Non-ocular AEs were the systemic events.
Time Frame: From baseline to Week 76
Population: Safety analysis population included all randomized participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Galegenimab Q4W | Galegenimab Q8W | All Sham
Number analyzed (Participants) | 149 | 75 | 148
percentage of participants | 57.7 | 54.7 | 62.8

5. Secondary Outcome: Percentage of Participants With Serious Adverse Events (SAEs)
Description: SAEs are defined as fatal, life threatening, requires or prolongs patient hospitalization, results in persistent or significant disability/incapacity, or is a significant medical event in the investigator's judgement.
Time Frame: From baseline to Week 76
Population: Safety analysis population included all randomized participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Galegenimab Q4W | Galegenimab Q8W | All Sham
Number analyzed (Participants) | 149 | 75 | 148
Percentage of Participants | 19.5 | 21.3 | 23

6. Secondary Outcome: Percentage of Participants With Adverse Events of Special Interest (AESIs)
Description: AESIs include 1.) cases of potential drug-induced liver injury that include an elevated alanine transaminase (ALT) or aspartate aminotransferase (AST) in combination with either an elevated bilirubin or clinical jaundice, as defined by Hy's Law 2.) Suspected transmission of an infectious agent by galegenimab 3.) AEs resulting from medication error 4.) Sight-threatening AEs of the following criteria: It causes a decrease of >= 30 letters in visual acuity (VA) score, compared with the most recent prior VA assessment, that lasts more than 1 hour and is attributable to galegenimab; it requires surgical intervention to prevent permanent loss of sight; associated with severe (Grade 4+) intraocular inflammation (IOI) and/or IOI-associated retinal vasculitis; in the opinion of the investigator, it may require medical intervention to prevent permanent loss of sight.
Time Frame: From baseline to Week 76
Population: Safety analysis population included all randomized participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Galegenimab Q4W | Galegenimab Q8W | All Sham
Number analyzed (Participants) | 149 | 75 | 148
Percentage of Participants | 6.7 | 6.7 | 2.0

7. Secondary Outcome: Percentage of Participants With Adverse Events Leading to Study Discontinuation
Description: as for outcome 4
Time Frame: From baseline to Week 76
Population: Safety analysis population included all randomized participants who received at least one dose of study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Galegenimab Q4W | Galegenimab Q8W | All Sham
Number analyzed (Participants) | 149 | 75 | 148
Percentage of Participants | 2.0 | 1.3 | 2.7

8. Secondary Outcome: Mean Change in Best Corrected Visual Acuity (BCVA) Score From Baseline to Week 72 as Assessed by Early Treatment Diabetic Retinopathy Study (ETDRS) Chart Under Low-luminance Conditions
Description: BCVA score was based on the number of letters read correctly on the ETDRS visual acuity chart assessed at a starting distance of 4 meters (m) under low-luminance conditions. A decrease in the VA score indicates a worsening in visual acuity. BCVA score testing was performed prior to dilating the eyes. BCVA score ranges from 0 to 100 letters in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). A negative change from baseline indicates a decrease in the visual acuity.
Time Frame: Baseline, Week 72
Population: mITT population includes all randomized patients who received at least one dose of study drug, and have a baseline measurement and at least one post-baseline measurement of GA area by FAF, subjects grouped according to treatment assigned at randomization. Participants analyzed in this outcome measure were those included in mixed models for repeated measures (MMRM) analysis.
Measure: Mean (Standard Error); unit: ETDRS letters
Arm/Group | Galegenimab Q4W | Galegenimab Q8W | All Sham
Number analyzed (Participants) | 138 | 67 | 132
ETDRS letters | -3.45 (1.344) | -3.54 (1.974) | -3.06 (1.339)
Statistical Analysis 1: Comparison: Galegenimab Q4W vs All Sham; Test type: Superiority; p = 0.8388, MMRM; Difference in Adjusted Means = -0.39, 95% CI 2-sided [-4.14 to 3.36], Standard Error of Mean 1.901
Statistical Analysis 2: Comparison: Galegenimab Q8W; Test type: Superiority; p = 0.8412, MMRM; Difference in Adjusted Means = -0.48, 95% CI 2-sided [-5.18 to 4.23], Standard Error of Mean 2.384

9. Secondary Outcome: Mean Change in BCVA Score From Baseline to Week 72 as Assessed by ETDRS Chart
Description: BCVA score was based on the number of letters read correctly on the ETDRS visual acuity chart assessed at a starting distance of 4 meters (m). A decrease in the VA score indicates a worsening in visual acuity. BCVA score testing was performed prior to dilating the eyes. BCVA score ranges from 0 to 100 letters in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). A negative change from baseline indicates a decrease in the visual acuity.
Time Frame: Baseline, Week 72
Population: as for outcome 8
Measure: Mean (Standard Error); unit: ETDRS letter
Arm/Group | Galegenimab Q4W | Galegenimab Q8W | All Sham
Number analyzed (Participants) | 138 | 67 | 132
ETDRS letter | -5.05 (1.444) | -5.68 (2.032) | -5.88 (1.456)
Statistical Analysis 1: Comparison: Galegenimab Q4W vs All Sham; Test type: Superiority; p = 0.6865, MMRM; Difference in Adjusted Means = 0.83, 95% CI 2-sided [-3.22 to 4.88], Standard Error of Mean 2.052
Statistical Analysis 2: Comparison: Galegenimab Q8W vs All Sham; Test type: Superiority; p = 0.9355, MMRM; Difference in Adjusted Means = 0.20, 95% CI [-4.73 to 5.13], Standard Error of Mean 2.500

ADVERSE EVENTS:
Time Frame: From baseline to Week 76
Description: Safety analysis population included all randomized participants who received at least one dose of study drug.
Arm/Group | Galegenimab Q4W | Galegenimab Q8W | All Sham
All-Cause Mortality (participants affected / at risk) | 5/149 | 1/75 | 4/148
Serious Adverse Events (participants affected / at risk) | 29/149 | 16/75 | 34/148
Other Adverse Events (participants affected / at risk) | 53/149 | 21/75 | 38/148
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Galegenimab Q4W (N=149) | Galegenimab Q8W (N=75) | All Sham (N=148)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (2) | 2 (3) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 2 (3)
Torsade de pointes (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Deafness unilateral (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Choroidal neovascularisation (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Iridocyclitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Macular hole (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Ocular hypertension (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal artery spasm (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinopathy proliferative (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Uveitis (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Vitritis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pancreatitis relapsing (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Tooth impacted (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 0 (0)
Swelling (General disorders) | 0 (0) | 0 (0) | 1 (1)
Swelling face (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumobilia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 3 (3) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Empyema (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Endophthalmitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Vascular graft infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Anaesthetic complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 3 (3)
Fracture displacement (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Blood sodium decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Intraocular pressure increased (Investigations) | 2 (4) | 0 (0) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 0 (0) | 1 (1)
Troponin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Desmoplastic melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Gastric cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Myoclonus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Device dislocation (Product Issues) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertensive urgency (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Galegenimab Q4W (N=149) | Galegenimab Q8W (N=75) | All Sham (N=148)
Conjunctival haemorrhage (Eye disorders) | 15 (19) | 6 (10) | 6 (9)
Posterior capsule opacification (Eye disorders) | 6 (8) | 3 (3) | 8 (9)
Retinal haemorrhage (Eye disorders) | 7 (8) | 5 (6) | 8 (14)
Vitreous detachment (Eye disorders) | 11 (12) | 3 (3) | 3 (4)
Vitreous floaters (Eye disorders) | 12 (12) | 3 (3) | 1 (1)
COVID-19 (Infections and infestations) | 10 (11) | 3 (3) | 10 (10)
Fall (Injury, poisoning and procedural complications) | 8 (9) | 1 (1) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-23): https://cdn.clinicaltrials.gov/large-docs/09/NCT03972709/Prot_SAP_001.pdf